CLINICAL TRIAL: NCT05377476
Title: Investigation of the Effects of Motor Imagery and Action Observation in People With Multiple Sclerosis
Brief Title: Effects of Motor Imagery and Action Observation in People With Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Collaborators: Bandırma Onyedi Eylül University (Other)
Responsible Party: Principal Investigator, Melike Sumeyye Ozen, Research Assistant, Bandırma Onyedi Eylül University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-5
Record Dates: First submitted 2022-05-12; First posted 2022-05-17 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Motor Imagery; Action Observation; Walking; Fatigue; Trunk Control
MeSH Terms: conditions — Multiple Sclerosis; Fatigue

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Motor Imagery Group (Experimental): Individuals included in this group will receive 20 minutes of motor imagery training in addition to 40 minutes of standard rehabilitation. Patients will be trained 3 days a week for 6 weeks.
  Interventions: Other: Motor Imagery training; Other: standard rehabilitation
- Action Observation Group (Experimental): Individuals included in this group will receive 20 minutes of action observation training in addition to 40 minutes of standard rehabilitation. Patients will be trained 3 days a week for 6 weeks.
  Interventions: Other: Action Observation training; Other: standard rehabilitation
- Control Group (Other): Individuals included in this group will receive only 40 minutes of standard rehabilitation. Patients will be trained 3 days a week for 6 weeks.
  Interventions: Other: standard rehabilitation

INTERVENTIONS:
Other: Motor Imagery training — Individuals included in this group will receive 20 minutes of motor imagery training in addition to 40 minutes of standard rehabilitation.
  Arms: Motor Imagery Group
Other: Action Observation training — Individuals included in this group will receive 20 minutes of action observation training in addition to 40 minutes of standard rehabilitation.
  Arms: Action Observation Group
Other: standard rehabilitation — 40 minutes of standard rehabilitation.

SUMMARY:
It was planned to examine the effects of motor imagery and action observation applied in addition to standard rehabilitation in people with multiple sclerosis on walking, fatigue, and trunk control.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-65
* A definitive diagnosis of MS by a neurologist according to the 2017 McDonald Criteria
* Expanded Disability Status Scale (EDSS) score of 4.0 and below (it is determined routinely by the physician during the examination)
* Not having an attack in the last 3 months
* A minimum score of 4 in each motor imagery ability (internal visual imagery, external visual imagery, and kinesthetic imagery) on the Movement Imagery Questionnaire-3 (MIQ-3)

Exclusion Criteria:

* cognitive impairment, defined as a Mini-Mental State Examination (MMSE) score of less than 24
* Having another musculoskeletal, cardiovascular, pulmonary, metabolic, or neurological disease severe enough to preclude participation in the study.
* Having severe vision and hearing problems

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
6 Min Walking Test | 6 week
  It will be used to measure walking distance. Before the test is administered, individuals will be given the necessary information and will be asked to walk as fast as possible on a 30-meter track for 6 minutes.

SECONDARY OUTCOMES:
Timed Up and Go Test | 6 week
  It will be used to evaluate the dynamic balance of individuals while walking. Individuals will be asked to stand up from the chair they are sitting on without support and walk a distance of 3 meters, then return from the designated area and sit on the chair without support.
Multiple Sclerosis Walking Scale-12 | 6 week
  It is a scale used to measure perceived walking ability. The lowest possible total score on the scale is "12," while the highest is "60". An increase in the total score indicates a negative impact on walking ability.
RehaGait® (Hasomed, Magdeburg, Germany) Gait Analysis | 6 week
  The device gives about the time-distance characteristics and kinematic data of the gait.
Fatigue Severity Scale | 6 week
  It is a scale that evaluates the extent to which fatigue affects the daily functions of MS patients. The lowest score that can be obtained from the scale is 7, while the highest score is 63. It is accepted that the severity of fatigue increases as the total score increases.
Trunk Impairment Scale | 6 week
  Trunk control was assessed using the Trunk Impairment Scale (TIS), which consists of three subscales: static sitting balance, dynamic sitting balance, and coordination. The lowest possible total score on the scale is "0", while the highest is "23". An increase in the total score indicates increased trunk control.

CONTACTS AND LOCATIONS:
Overall Officials: Melike Sumeyye Ozen, M.Sc., Principal Investigator — Bandırma Onyedi Eylül University
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No